CLINICAL TRIAL: NCT05530707
Title: Avaliação de Aceitabilidade dérmica, eficácia Hidratante, restauração da Barreira e equilíbrio da Microbiota da Pele atópica de um Produto Hidratante - Estudo Clínico, Instrumental e Subjetivo.
Brief Title: Evaluation of Acceptability, Skin Barrier Restoration and Balance of Atopic Skin Using Moisturizer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farmoquimica S.A. (Industry)
Collaborators: Medcin Instituto da Pele (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EN21-0556-01_EN22-2004-01
Record Dates: First submitted 2022-08-11; First posted 2022-09-07 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Atopic Dermatitis
Keywords: cosmetics
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microbiome (Experimental): 13 participants using the product for 30 days. Aims to evaluate the quantification of S. Aureus in the skin before and after usage.
  Interventions: Other: Moisturizer containing saccharide isomerate and niacinamide
- Clinical Trial (Experimental): 36 participants using the product for 60 days. Aims to evaluate the clinical, subjective and instrumental usage.
  Interventions: Other: Moisturizer containing saccharide isomerate and niacinamide

INTERVENTIONS:
Other: Moisturizer containing saccharide isomerate and niacinamide — Moisturizer containing saccharide isomerate and niacinamide

SUMMARY:
A unicentric, blind, non-comparative clinical study to evaluate the efficacy of a moisturizer in reducing clinical symptons of atopic dermatites in children through clinical, subjective and instrumental evaluations.

DETAILED DESCRIPTION:
A unicentric, blind, non-comparative clinical study to evaluate the efficacy of a moisturizer in reducing clinical symptons of atopic skin dermatites in children through clinical, subjective and instrumental evaluations.

Participants will be divided into 2 groups - (Group 1) Microbiome analysis; and (Group 2) Acceptabily and efficacy

Group 1: It will be necessary 13 participants aged between 05 and 12 years old with historical of atopia

The participant will remain in the study for 30 days using the product. Visits will be scheduled in D0 and D30. On both visits, samples will be collect to quantify Staphylococcus aureus using qPCR

Group 2: It will be necessary 36 participants aged between 05 and 12 years old with historical of atopia

The participant will remain in the study for 60 days using the product. Visits will be scheduled in D0, D7, D30 and D60.

Instrumental evaluations: It will be evaluate on each visit:

Skin hidration using Corneometer - D0, D7, D30, D60 Transepidermic water loss using TEWL - D0, D7, D30, D60 Skin barrier restoration using Confocal Microscopy - D0, D30, D60

Participants will respond to a subjective assessment using a questionnaire to capture possible feelings of discomfort during the study e subjective efficiency.

A dermatologist will be available to monitor the participants throughout the study and respond a assessment of clinical efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and consent to participation in this clinical trial, manifested through the signatures of the Informed Consent (TCLE) by at least one of the minor's legal guardians, and signature of the Free and Informed Consent Term (TALE) by the minor, when applicable (≥07 years);
2. Agreement to participate the procedures and requirements of the study and attend the Institute on the day(s) and time(s) determined for the assessments accompanied by the responsible
3. Participants with a history of atopy
4. Participants with presence of dry skin with dryness, flaking and mild itching in the pretibial region
5. Presence of active lesions of atopic dermatitis in the cubital cavus region for group 1 of participants who did not need other topical treatments besides the moisturizer

Exclusion Criteria:

1. Pregnancy/lactation or intention to become pregnant during the study period;
2. Presence of active lesions of atopic dermatitis for group 2 of participants - Clinical study;
3. Use of the following topical or systemic medications: immunosuppressants, antihistamines, anti-inflammatory drugs corticosteroids up to 30 days prior to selection. For immunosuppressants, the interval should be 3 months prior to selection;
4. Presenting or having a history of other concomitant skin conditions (e.g., psoriasis or lupus erythemasus) that interferes with the evaluations of the effect of the investigational product of the study on AD;
5. Participants currently presenting a skin infection requiring treatment or are currently in need of treatment with topical or systemic antibiotics;
6. Any serious concomitant disease in which the need for the use of systemic corticosteroids is expected or which, otherwise interfere with study participation or require frequent active monitoring (e.g., asthma chronicunstable);
7. Unable or unwilling to be available throughout the study and/or not be willing to follow the study restrictions/procedures;
8. Stomach diseases such as gastritis and ulcers;
9. Chronic use of corticosteroids (systemic or topical);
10. Chronic kidney diseases, chronic liver diseases;
11. Clinical evidence of immunosuppression;
12. Allergic history of category products;
13. Participants with known congenital or acquired immunodeficiency;
14. Relevant clinical history or current evidence of alcohol or other drug abuse;
15. known history or suspected intolerance of products of the same category;
16. Intense sun exposure up to 30 days before evaluation;
17. Professionals directly involved in the present study;
18. Other conditions considered by the evaluating physician as reasonable for disqualification from the participation of the study. If yes, it should be described under observation in the clinical file.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Acceptability in real conditions of use by questionnaire | Day 60
  Confirm in real conditions of use, the absence of risk and irritation and capture feelings of discomfort in the population studied (0 meaning no risk).
Change of qPCR quantification of Staphylococcus aureus | Change from Baseline (Day 0) and day 30
  Evaluate the change in the skin microbiota by quantification of qPCR of Staphylococcus aureus in the skin before (D0) and after 30 (D30) days of continuous use of the product.

SECONDARY OUTCOMES:
Clinical Evaluation through dermatological questionnaire | Day 60
  Evaluate the efficacy in reducing the signs of atopic dermatitis through dermatological clinical evaluation after 60 days of continuous use of the product
Increase of skin hidration using instrumental evaluation - Corneometer | Day 0, 7, 30 and 60
  Evaluate the moisturizing efficacy immediately (D0) after application of the investigational product and after 7 (D7), 30 (D30) and 60 (D60) days of continuous use, through the Corneometer equipment®
Evaluation of recovery of skin barrier through instrumental method - TEWL | Day 7, 30 and 60
  Evaluate the efficacy in the recovery of the skin barrier after 7 (D7), 30 (D30) and 60 (D60) days of continuous use of the product through the Tewameter equipment®
Strengthening of the skin barrier | Day 0, 30 and 60
  Evaluate the strengthening of the skin barrier in D0 and after 30 (D30) and 60 (D60) days of continuous use of the product by confocal reflectance microscopy
Subjective efficacy from the participants | Day 0, 7, 30 and 60
  Evaluate the perceived efficacy of the product from the participant's point of view through a subjective questionnaire immediately after the first application (Timed) and after 7 (D7), 30 (D30) and 60 (D60) days of continuous use of the product
Improvement of Quality of Life | Day 0, 7, 30 and 60
  Evaluate the improvement of the quality of life of the atopic dermatitis carrier through a questionnaire on quality of life in D0 and after 30 and 60 days of continuous use of the product

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele, Osasco, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: D60